CLINICAL TRIAL: NCT00053703
Title: Treatment of Schizophrenia and Related Disorders in Children and Adolescents
Brief Title: Treatment of Early Onset Schizophrenia Spectrum Disorders (TEOSS)
Acronym: TEOSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01 MH 615218-01A; U01MH062726 (NIH); U01MH061355-01A1 (NIH); U01MH062726-01 (NIH); U01MH061464-01A1 (NIH); NCT00030251 (obsolete NCT alias); NCT00043290 (obsolete NCT alias)
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
Keywords: Psychotic Disorders; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Olanzapine; Molindone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- olanzapine (Active Comparator): oral olanzapine 5-20mg per day for up to 52 weeks
  Interventions: Drug: Olanzapine (enrollment closed in this treatment)
- risperidone (Active Comparator): oral risperidone 0.5mg to 6mg daily for up to 52 weeks
  Interventions: Drug: Risperidone
- molindone (Active Comparator): oral molindone from 10-140mg/daily for up to 52 weeks
  Interventions: Drug: Molindone

INTERVENTIONS:
Drug: Risperidone — oral risperidone 0.5mg to 6mg daily for up to 52 weeks
  Other Names: Risperdal
  Arms: risperidone
Drug: Olanzapine (enrollment closed in this treatment) — oral olanzapine 5-20mg per day for up to 52 weeks
  Other Names: Zyprexa
  Arms: olanzapine
Drug: Molindone — oral molindone from 10-140mg/daily for up to 52 weeks
  Other Names: Moban
  Arms: molindone

SUMMARY:
This study will evaluate the safety and efficacy of risperidone (Risperdal®), olanzapine (Zyprexa®), and molindone (Moban®) for the treatment of children and adolescents with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Little research has been conducted on the use of psychotropic agents in children and adolescents with early onset schizophrenia spectrum disorders. This study will compare antipsychotic agents with different mechanisms of action in children and adolescents who have schizophrenia or schizoaffective disorder with active psychotic symptoms.

Participants are randomly assigned to receive risperidone (Risperdal), olanzapine (Zyprexa), or molindone (Moban) for 8 weeks. After 11/2005, no additional patients will be assigned to olanzapine treatment. Patients with significant improvement and without side effects continue maintenance therapy for another 44 weeks. Participants who show significant negative symptoms after 8 weeks may be started on a mood stabilizer or antidepressant. Weight gain, metabolic changes, neurocognition, functional outcome, psychotic symptoms, extrapyramidal side effects, and the ability to sustain effective therapy over time are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, schizophreniform disorder, or schizoaffective disorder with psychotic symptoms
* Free of depot antipsychotic medication for at least 6 months. Oral antipsychotic medication at entry into the study is allowed, provided the participant has not had an adequate trial during the present episode of psychosis.
* If taking antidepressant or mood stabilizing medication, stable dosing for at least 30 days prior to entry.
* Good physical health

Exclusion Criteria:

* Risperidone (RIS), olanzapine (OLA)*, or molindone (MOL) for 8 weeks or more during THIS episode, with 2 weeks at the maximal dose (6 mg/day of RIS, 20 mg/day of OLA, or 140 mg/day of MOL)
* If using antidepressant and/or mood stabilizing medications, treatment for fewer than 30 days immediately before entry
* Intolerance or nonresponse to RIS, OLA*, or MOL during any previous treatment
* Bipolar affective disorder,post traumatic stress disorder, personality disorder, or psychosis not otherwise specified
* Currently meeting Diagnostic and Statistical Manual version IV (DSM IV) criteria for major depression episode
* DSM IV criteria for substance abuse or dependence with intention to continue illicit substance abuse
* Endocrinological or neurological conditions which confound the diagnosis or are a contraindication to treatment with antipsychotics
* Mental retardation
* Risk of suicide or homicide that is not adequately controlled in the current setting
* Pregnancy or refusal to practice contraception during the study

"*" OLA exclusion not applicable after 11/2005

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2002-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, M.D., Study Chair — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Cambridge Health Alliance, Medford, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] McCLELLAN J, Sikich L, Findling RL, Frazier JA, Vitiello B, Hlastala SA, Williams E, Ambler D, Hunt-Harrison T, Maloney AE, Ritz L, Anderson R, Hamer RM, Lieberman JA. Treatment of early-onset schizophrenia spectrum disorders (TEOSS): rationale, design, and methods. J Am Acad Child Adolesc Psychiatry. 2007 Aug;46(8):969-978. doi: 10.1097/CHI.0b013e3180691779. PMID 17667476
- [Result] Frazier JA, McCLELLAN J, Findling RL, Vitiello B, Anderson R, Zablotsky B, Williams E, McNAMARA NK, Jackson JA, Ritz L, Hlastala SA, Pierson L, Varley JA, Puglia M, Maloney AE, Ambler D, Hunt-Harrison T, Hamer RM, Noyes N, Lieberman JA, Sikich L. Treatment of early-onset schizophrenia spectrum disorders (TEOSS): demographic and clinical characteristics. J Am Acad Child Adolesc Psychiatry. 2007 Aug;46(8):979-988. doi: 10.1097/chi.0b013e31807083fd. PMID 17667477
- [Result] Findling RL, Johnson JL, McClellan J, Frazier JA, Vitiello B, Hamer RM, Lieberman JA, Ritz L, McNamara NK, Lingler J, Hlastala S, Pierson L, Puglia M, Maloney AE, Kaufman EM, Noyes N, Sikich L. Double-blind maintenance safety and effectiveness findings from the Treatment of Early-Onset Schizophrenia Spectrum (TEOSS) study. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):583-94; quiz 632. doi: 10.1016/j.jaac.2010.03.013. Epub 2010 May 1. PMID 20494268
- [Derived] Taylor JH, Appel S, Eli M, Alexander-Bloch A, Maayan L, Gur RE, Bloch MH. Time to Clinical Response in the Treatment of Early Onset Schizophrenia Spectrum Disorders Study. J Child Adolesc Psychopharmacol. 2021 Feb;31(1):46-52. doi: 10.1089/cap.2020.0030. Epub 2020 Jul 1. PMID 32633541
- [Derived] Taylor JH, Jakubovski E, Gabriel D, Bloch MH. Predictors and Moderators of Antipsychotic-Related Weight Gain in the Treatment of Early-Onset Schizophrenia Spectrum Disorders Study. J Child Adolesc Psychopharmacol. 2018 Sep;28(7):474-484. doi: 10.1089/cap.2017.0147. Epub 2018 Jun 19. PMID 29920116
- [Derived] Gabriel D, Jakubovski E, Taylor JH, Artukoglu BB, Bloch MH. Predictors of treatment response and drop out in the Treatment of Early-Onset Schizophrenia Spectrum Disorders (TEOSS) study. Psychiatry Res. 2017 Sep;255:248-255. doi: 10.1016/j.psychres.2017.05.038. Epub 2017 May 30. PMID 28595147
- [Derived] Frazier JA, Giuliano AJ, Johnson JL, Yakutis L, Youngstrom EA, Breiger D, Sikich L, Findling RL, McClellan J, Hamer RM, Vitiello B, Lieberman JA, Hooper SR. Neurocognitive outcomes in the Treatment of Early-Onset Schizophrenia Spectrum Disorders study. J Am Acad Child Adolesc Psychiatry. 2012 May;51(5):496-505. doi: 10.1016/j.jaac.2012.02.001. Epub 2012 Mar 13. PMID 22525956
- [Derived] Sikich L, Frazier JA, McClellan J, Findling RL, Vitiello B, Ritz L, Ambler D, Puglia M, Maloney AE, Michael E, De Jong S, Slifka K, Noyes N, Hlastala S, Pierson L, McNamara NK, Delporto-Bedoya D, Anderson R, Hamer RM, Lieberman JA. Double-blind comparison of first- and second-generation antipsychotics in early-onset schizophrenia and schizo-affective disorder: findings from the treatment of early-onset schizophrenia spectrum disorders (TEOSS) study. Am J Psychiatry. 2008 Nov;165(11):1420-31. doi: 10.1176/appi.ajp.2008.08050756. Epub 2008 Sep 15. PMID 18794207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2002 to May 2006, youth were screened at four academic sites: University of North Carolina at Chapel Hill, McLean Hospital and Cambridge Health Alliance at Harvard Medical School, University of Washington, and Case Western Reserve University.
Period: Overall Study
Arm/Group | Olanzapine | Risperidone | Molindone
Started | 35 | 41 | 40
Completed | 17 | 28 | 25
Not Completed | 18 | 13 | 15

BASELINE CHARACTERISTICS:
Population: We are referring to the population of participants who had baseline assessment, took at least one dose of trial medication, and had at least one post-baseline assessment. There were 3 randomized subjects, on in each treatment group, who did not take at least one dose of study medication and are not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Risperidone | Molindone | Total
Number analyzed (Participants) | 35 | 41 | 40 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 40 | 39 | 114
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.84 (2.41) | 14.54 (2.38) | 14.3 (2.4) | 14.25 (2.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 17 | 41
  Male | 25 | 27 | 23 | 75
Region of Enrollment [Number; unit: participants]
  United States | 35 | 41 | 40 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at 8 Weeks
Description: Assessed with the Positive and Negative Syndrome Scale in which a clinician rates various psychotic symptoms on the basis of observation of the participant, interview with the participant, and review of all other available information including informant reports. The scale consists of 30 items which are rated categorically between 1 - no symptoms to 7 - extreme symptoms. The minimal score is 0 and the maximal score is 210, with higher scores reflecting more symptoms. Typically scores > that 60 are considered clinically significant.
Time Frame: 8 weeks
Population: All randomized patients who took at least one dose of drug and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
units on a scale | -26.6 (17.8) | -23.7 (25.5) | -27.0 (17.7)
Statistical Analysis 1: Comparison: Olanzapine vs Risperidone vs Molindone; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Weight at Week 8
Description: change in weight from baseline to week 8 in kg
Time Frame: 8 weeks
Population: All randomized patients who took at least one dose of drug and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
Kg | 6.12 (3.60) | 3.64 (3.95) | 0.34 (2.86)

3. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale at Week 8
Description: Barnes Akathisia Scale is a clinician rated scale which considers information based on observation of the participant as well as participant report. The scale includes 3 items rated between 0- none to 3 severe and 1 summary item rated between 0 none to 5 severe. All items are summed to obtain the total score. The minimal total score is 0 and the maximal score is 14 with higher scores reflecting more severe akathisia. A score of 4 or more is clinically significant.
Time Frame: 8 weeks
Population: All randomized patients who took at least one dose of drug and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
units on a scale | 0.19 (2.12) | 0.41 (2.37) | 1.23 (3.34)

4. Primary Outcome: Change From Baseline in PANSS Positive Symptom Subscale Score at 8 Weeks.
Description: The PANSS (described above) includes 7 items that reflect positive psychotic symptoms such as hallucinations and delusions. As are all items within the PANSS, items are categorically rated by the clinician between 0 - no symptoms to 7 extreme symptoms. The minimal score is 0 reflecting no positive symptoms to 49 reflecting that all items were extreme. Higher scores reflect more severe symptoms. Scores above 18 are usually clinically significant.
Time Frame: 8 weeks
Population: All randomized patients who took at least one dose of drug and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
units on a scale | -8.9 (6.0) | -8.4 (8.1) | -8.8 (5.4)

5. Primary Outcome: Change From Baseline in PANSS Negative Symptom Subscale at Week 8
Description: The PANSS (described above) includes 7 items that reflect negative psychotic symptoms such as amotivation and social withdrawal. As are all items within the PANSS, items are categorically rated by the clinician between 0 - no symptoms to 7 extreme symptoms. The minimal score is 0 reflecting no positive symptoms to 49 reflecting that all items were extreme. Higher scores reflect more severe symptoms. Scores above 18 are usually clinically significant.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
units on a scale | -5.3 (7.6) | -5.1 (7.8) | -5.8 (6.8)

6. Secondary Outcome: Change From Baseline in Body Mass Index Change, kg/m2, at Week 8
Description: Change from baseline in Body Mass Index Change, kg/m2, at week 8, last observation was carried forward for individuals who withdrew from treatment early.
Time Frame: 8 weeks
Population: All randomized patients who took at least one dose of drug and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Olanzapine | Risperidone | Molindone
Number analyzed (Participants) | 35 | 41 | 40
kg/m2 | 1.27 (1.51) | 2.20 (1.24) | 0.15 (1.26)

ADVERSE EVENTS:
Time Frame: 8 weeks, Systematic events
Arm/Group | Olanzapine | Risperidone | Molindone
Serious Adverse Events (participants affected / at risk) | 2/35 | 4/41 | 2/40
Other Adverse Events (participants affected / at risk) | 26/35 | 35/41 | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=35) | Risperidone (N=41) | Molindone (N=40)
Psychiatric Hospitalization (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1)
Suicidal Thoughts (life-threatening) (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=35) | Risperidone (N=41) | Molindone (N=40)
Agitation (Psychiatric disorders) | 6 (6) | 5 (5) | 7 (7)
Akathisia (Nervous system disorders) | 5 (5) | 4 (4) | 17 (17)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3) | 9 (9)
Blurred Vision (Eye disorders) | 0 (0) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7) | 1 (1)
Depression (Psychiatric disorders) | 6 (6) | 5 (5) | 4 (4)
Dystonia (Nervous system disorders) | 6 (6) | 5 (5) | 1 (1)
Increase in appetite (General disorders) | 14 (14) | 7 (7) | 3 (3)
Insomnia (General disorders) | 2 (2) | 6 (6) | 6 (6)
Irritability (Psychiatric disorders) | 9 (9) | 8 (8) | 9 (9)
Menstrual Irregularities (General disorders) | 1 (1) | 2 (2) | 2 (2)
Sedation/Drowsiness (General disorders) | 11 (11) | 13 (13) | 16 (16)
weight gain (General disorders) | 17 (17) | 7 (7) | 3 (3)

LIMITATIONS AND CAVEATS:
The most significant weakness of this study was the sample size, which was sufficient only to detect large differences across the three treatments and limited our ability to identify predictors of response or adverse effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No